CLINICAL TRIAL: NCT01816789
Title: Age Versus Ovarian Reserve Markers Based Therapy in IN Vitro Fertilization
Brief Title: Age Versus Ovarian Reserve Markers Based Therapy in IVF (IVF)/Intracytoplasmic Sperm Injection (ICSI) Cycles
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Optimal response: 63% nomogram, 42% controls, overcoming the stopping rule for interim analysis
Sponsor: Andros Day Surgery Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANDROS-01-13
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: In Vitro Fertilization; Ovarian Stimulation
Keywords: Starting dose; rFSH; controlled; ovarian; stimulation; IVF/ICSI; cycles
MeSH Terms: interventions — Buserelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: "age" (Active Comparator): Group A: long standard protocol (buserelin 0.1 ml s.c. twice per day from the 21st day of the cycle, until the end of gonadotropin administration) + 150 IU of rFSH (starting dose) if female age was ≤35 years or 225 IU of rFSH if female age was ≥ 36 years.
  Interventions: Drug: rFSH; Drug: buserelin
- Group B: "nomogram" (Experimental): Group B: long standard protocol (buserelin 0.1 ml s.c. twice per day from the 21st day of the cycle until the end of gonadotropin administration) + individualized starting dose of rFSH on the basis of the nomogram.
  Interventions: Drug: rFSH; Drug: buserelin

INTERVENTIONS:
Drug: rFSH
Drug: buserelin

SUMMARY:
This randomized controlled trial has been designed for carrying out a comparison of new AMH (Anti-Müllerian Hormone)-based individualized treatment (using a nomogram) with the wide accepted age-based strategy. The main objective of the trial is to assess whether an individualized FSH starting dose can increase the rate of women with an adequate ovarian response in terms of retrieved oocytes (optimal number of retrieved oocytes: 8-14).

DETAILED DESCRIPTION:
Before clinicians can adopt any model into routine clinical practice, the accuracy of the model should be independently evaluated in a population different from the one on which the model was elaborated. External validation of the model is therefore crucial to assess the generalizability to other populations.

In the present RCT the new AMH-based individualized treatment will be compared to the wide accepted age-based strategy.

Primary endpoint:

The percentage of women with an appropriate number (n=8-14) of retrieved oocytes in IVF/ICSI cycle.

Secondary endpoints:

1. Serum E2 levels on r-hCG day
2. Serum P levels on r-hCG day
3. Number of growing follicles (≥11mm) on r-hCG day
4. Number of large (≥ 17 mm) ovarian follicles on r-hCG day
5. Total r-FSH dose employed
6. Treatment duration
7. Rate of women with dose adjustment
8. Number of cancelled cycles because of poor and hyper-response
9. Fertilization rate
10. Embryos obtained
11. Implantation rates
12. Biochemical pregnancy rates
13. Clinical pregnancy rates
14. OHSS rates

ELIGIBILITY:
Inclusion Criteria:

* first or second IVF/ICSI attempt (the second one after 6 months from the first one);regular menstrual cycles (25-33 days);female age ≤ 40; day 3 FSH ≤ 15IU/L;treatment with a long GnRH agonist protocol (buserelin)+rFSH;BMI: >18 and ≤ 25 kg/m2;presence of both ovaries.

Exclusion Criteria:

* irregular cycles, anovulatory infertility, endometriosis III-IV stage AFS, use of adjunctive therapies for stimulation, evidence of PCO status, previous ovarian surgery, presence of ovarian cysts, history of PID, use of hormonal contraception in the previous 3 months, any known metabolic or endocrinological disease, AMH levels < 1 and > 4.0 ng/ml

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The percentage of women with an appropriate number (N=8-14) of retrieved oocytes in IVF/ICSI cycles | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- ANDROS Day Surgery Clinic, Palermo, Sicily, Italy